CLINICAL TRIAL: NCT06651762
Title: Ultra Sound Guided Genicular Nerves Cooled Radiofrequency Ablation in Total Knee Replacement Surgeries
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: FMASU R221/2024
Record Dates: First submitted 2024-10-19; First posted 2024-10-22 (Actual); Last update posted 2025-02-24 (Actual); Status verified 2024-09

CONDITIONS: Osteoarthritis of Knee
MeSH Terms: conditions — Osteoarthritis, Knee | interventions — Injections, Epidural

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- lumber epidural anesthesia (Experimental): Patients will receive epidural anesthesia intra operative
  Interventions: Procedure: Epidural
- lumber Epidural and unilateral genicular nerve ablation: (Experimental): Patient will receive lumber epidural anesthesia and unilateral genicular nerve cooled radio frequency ablation pre-operative
  Interventions: Procedure: unilateral Radiofrequency; Procedure: Epidural
- Epidural and bilateral genicular nerve ablation (Experimental): Patient will receive lumber epidural anesthesia and bilateral genicular nerve cooled radio frequency ablation pre-operative
  Interventions: Procedure: bilateral Radiofrequency; Procedure: Epidural

INTERVENTIONS:
Procedure: unilateral Radiofrequency — unilateral genicular nerve cooled radio frequency ablation pre-operative
  Arms: lumber Epidural and unilateral genicular nerve ablation:
Procedure: bilateral Radiofrequency — bilateral genicular nerve cooled radio frequency ablation pre-operative
  Arms: Epidural and bilateral genicular nerve ablation
Procedure: Epidural — Patients will receive epidural anesthesia intra operative and epidural analgesia post-operative

SUMMARY:
Total Knee Replacement surgery is common procedure that is usually done for patients suffering from persistent pain with limitation of movement. Unfortunately, they do suffer after the operation as it is associated still with significant pain that affect the rehabilitation plan, hospital length of stay, life style and patient satisfaction. New approaches are rising every day to add to the multimodal management plan. Genicular nerves cooled radiofrequency ablation is a new approach that can be simply done U.S. guided with little side effects, if any, and great results.

DETAILED DESCRIPTION:
the study measures the efficacy of genicular nerves cooled radiofrequency ablation in enhancing quality of rehabilitation in patients undergoing total knee replacement

ELIGIBILITY:
Inclusion Criteria:• Undergoing a scheduled unilateral total knee replacement surgery

-

Exclusion Criteria:

* • Allergy to any of the drugs used in the study

  * Alcohol or drug abuse
  * Psychiatric disease

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Estimated)
Dates: Start 2024-10-14 (Actual); Primary Completion 2025-04-13 (Estimated); Study Completion 2025-06-13 (Estimated)

PRIMARY OUTCOMES:
o Epidural rescue doses | 1st 48 hours
  rescue doses reflects degree of pain control

CONTACTS AND LOCATIONS:
Locations (1):
- faculty of medicine Ain Shams University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Yes
Data required for interpretation of results will be shared
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: 6 months to 12 months after publication